CLINICAL TRIAL: NCT03995043
Title: Project for Reproductive Equity Through Volunteers and Entrepreneurship, Networks and Technology: The PREVENT Project Protocol
Brief Title: Project for Reproductive Equity Through Volunteers and Entrepreneurship, Networks and Technology
Acronym: PREVENT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Karen Yeates (Other)
Responsible Party: Sponsor-Investigator, Dr. Karen Yeates, Principal Investigator, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: ST-POC-1807-15184
Record Dates: First submitted 2019-06-13; First posted 2019-06-21 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Contraception; Pregnancy Related; Reproductive Behavior
MeSH Terms: conditions — Reproductive Behavior | interventions — Educational Status; Health Services Accessibility

STUDY DESIGN:
Intervention Model Description: This is an individually randomized parallel group study design.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants are blinded through the study arm and the outcomes assessor and investigator are blinded to participant group assignment for the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Intervention (Experimental): 1. Education about contraceptive use, reproductive health and family planning services through SMS messages on SRH.
  2. Personal Support from community peer mentor to access counselling services through SRH
  Interventions: Behavioral: Education; Behavioral: Personal Support
- Case Intervention (Experimental): 1. Education about contraceptive use, reproductive health and family planning services through SMS messages on SRH.
  2. Personal Support from community peer mentor to access counselling services through SRH
  3. Access to Contraception and counselling and service provision will be provided by the mobile reproductive health team at contraceptive access points.
  Interventions: Behavioral: Education; Behavioral: Personal Support; Behavioral: Access to contraception

INTERVENTIONS:
Behavioral: Education — Receive educational SMS (text) messages about contraceptive use and family planning on SRH and access individually tailored educational resources through interactive voice response (IVR) services/system via PREVENT mobile platform.
Behavioral: Personal Support — Contact with a female business owner within the community (hair saloons, tailors, female clothing stores) act as both a confidential, and non-judgmental resource to answer questions and provide counselling in SRH to study participants.
Behavioral: Access to contraception — Will be provided by the mobile reproductive health team at contraceptive access points, and, at the health facility partners who will be providing full reproductive health services to program participants and will be the access points for Intra-Uterine Device (IUD) insertion where requested and medically suitable. Results of point of care urine HCG (pregnancy) testing (voluntary at enrollment and mandatory when accessing contraceptive services)
  Arms: Case Intervention

SUMMARY:
The PREVENT Project is a multifaceted, adolescent friendly, culturally competent program aimed to address the issues surrounding unplanned pregnancies and lack of access and uptake of contraceptive services among adolescent girls. The intervention uses a mobile platform that provides educational SMS (Short Message Service) messaging, interactive voice response, and connects adolescent girls to community based AFSRH (Adolescent Friendly Sexual Reproductive Health) counselling services, as well as discreet contraceptive access points headed by female entrepreneurs. The program will be piloted for 12 months in various wards and villages in rural and urban Kilimanjaro, Tanzania.The acceptability and practicality of the intervention will be assessed using mixed methods. Questionnaires and focus groups will be conducted with the study participants, as well as the medical and non-medical volunteers at the start and end of the pilot. The study will be heavily supported by all-female non-medical social entrepreneurs and sexual reproductive health community mentors (volunteers), and, all-female medical reproductive health team. Recruitment will also take place in hair saloons (local hair braiding and styling establishments) and other female run business such as tailors and female clothing stores that have enlisted to become contraceptive access points in the study. There will be 2 intervention groups, control and case group. Both groups will receive educational SMS (text) messages on SRH (Sexual Reproductive Health) and access individually tailored educational resources through interactive voice response (IVR) services/system via PREVENT mobile platform. In addition to personal support to be able to contact with a SRH community peer mentor in the community for AFSRH counselling and support. The case group will then have access to contraception provided with detailed and discreet information on accessing PREVENT contraceptive access points in all communities included in the study.

DETAILED DESCRIPTION:
The PREVENT study seeks to impact knowledge, perceptions, and behavioural changes regarding SRH among adolescent girls. As a result, the data collected in the PREVENT study will be grouped into two main themes: SRH knowledge and attitudes, as well as family planning (pregnancy avoidance) and contraceptive services uptake and outcomes. All data collected during the study will be directly entered and stored into the secure PREVENT mobile platform and related secure storage functions within the platform.

ELIGIBILITY:
Inclusion Criteria:

* Women 15-19 years of age
* Reside within the study area for the duration of the study
* Have a personal mobile phone and be willing to provide the phone number to the researchers to receive the intervention messages
* Report being SMS literate (ie. able to read text messages in English or Swahili)
* Be able and willing to return for follow-up after 12 months
* Be able and willing to give written informed consent for enrollment in the study

Exclusion Criteria:

* Be pregnant or planning pregnancy within 12 months (assessed when obtaining consent using HCG (human chorionic gonadotropin) urine dipstick).
* Participation in another study or intervention that may affect the outcome of this study
* Already utilizing a long-term form of contraception such as intra-uterine device, or implantable or inject-able contraception
* Having a non-medical condition detected through screening that hinders study participation such as developmental or cognitive delay

Ages: 15 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Study dealing with female contraception use and access.
Enrollment: 198 (Estimated)
Dates: Start 2026-12 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in unmet need for contraceptives at 6 months | 6 month
  Percent change in unmet need for contraceptives among study participants using Tanzania Demographic and health survey.
Change in unmet need for contraceptives at 12 months | 12 month
  Percent change in unmet need for contraceptives among study participants using Tanzania Demographic and health survey.

SECONDARY OUTCOMES:
Questionnaire to test knowledge regarding sexual and reproductive health | 12 month post randomization
  Change in health knowledge by participants regarding sexual and reproductive health through engagement with the program using the Family Health International/Pathfinder adolescent fertility questionnaires. Focused on sociodemographic characteristics, levels of sexual activity, knowledge and use of contraceptives, incidence and outcomes of pregnancy, and knowledge and sources of information on reproductive health topics.
Change in the number of pregnancies among women at 6 months | 6 month post randomization
  Change in unwanted/unplanned pregnancies among participants in the program
Change in the number of pregnancies among women at 12 months | 12 month post randomization
  Change in unwanted/unplanned pregnancies among participants in the program

OTHER OUTCOMES:
Number of participants to use voice response and access counseling | 12 months post randomization
  Number of beneficiaries who utilize the interactive voice response system and access AFSRH counseling

CONTACTS AND LOCATIONS:
Locations (1):
- Queens University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ministry of Health, Community Development, Gender, Elderly and Children (TZ). Tanzania Demographic and Health Survey and Malaria Indicator Survey (TDHS-MIS) 2015-16 [Internet]. Dar es Salaam: Ministry of Health, Community Development, Gender, Elderly and Children, 2016 [cited 2018 Sept. 19]. 591 p. Available from: https://dhsprogram.com/publications/publication-fr321-dhs-final-reports.cfm
- [Background] Ministry of Health, Community Development, Gender, Elderly and Children (TZ). The National Road Map Strategic Plan to Improve Reproductive, Maternal, Newborn, Child & Adolescent Health in Tanzania (2016-2020) [Internet]. Dar es Salaam: Ministry of Health, Community Development, Gender, Elderly and Children, 2016 [cited 2018 Sept. 19]. 132 p. Available from: https://www.globalfinancingfacility.org/national-road-map-strategic-plan-improve-reproductive-maternal-newborn-child-adolescent-health
- [Background] Rusibamayila A, Phillips J, Kalollela A, Jackson E, Baynes C. Factors influencing pregnancy intentions and contraceptive use: an exploration of the 'unmet need for family planning' in Tanzania. Cult Health Sex. 2017 Jan;19(1):1-16. doi: 10.1080/13691058.2016.1187768. Epub 2016 Jun 14. PMID 27297661
- [Background] Sweya MN, Msuya SE, Mahande MJ, Manongi R. Contraceptive knowledge, sexual behavior, and factors associated with contraceptive use among female undergraduate university students in Kilimanjaro region in Tanzania. Adolesc Health Med Ther. 2016 Oct 3;7:109-115. doi: 10.2147/AHMT.S108531. eCollection 2016. PMID 27757057
- [Background] Sedekia Y, Jones C, Nathan R, Schellenberg J, Marchant T. Using contraceptives to delay first birth: a qualitative study of individual, community and health provider perceptions in southern Tanzania. BMC Public Health. 2017 Oct 3;17(1):768. doi: 10.1186/s12889-017-4759-9. PMID 28974208
- [Background] Kabagenyi A, Reid A, Ntozi J, Atuyambe L. Socio-cultural inhibitors to use of modern contraceptive techniques in rural Uganda: a qualitative study. Pan Afr Med J. 2016 Oct 17;25:78. doi: 10.11604/pamj.2016.25.78.6613. eCollection 2016. PMID 28292041
- [Background] Haslegrave M. Ensuring the inclusion of sexual and reproductive health and rights under a sustainable development goal on health in the post-2015 human rights framework for development. Reprod Health Matters. 2013 Nov;21(42):61-73. doi: 10.1016/S0968-8080(13)42742-8. PMID 24315064
- [Background] Patton GC, Sawyer SM, Santelli JS, Ross DA, Afifi R, Allen NB, Arora M, Azzopardi P, Baldwin W, Bonell C, Kakuma R, Kennedy E, Mahon J, McGovern T, Mokdad AH, Patel V, Petroni S, Reavley N, Taiwo K, Waldfogel J, Wickremarathne D, Barroso C, Bhutta Z, Fatusi AO, Mattoo A, Diers J, Fang J, Ferguson J, Ssewamala F, Viner RM. Our future: a Lancet commission on adolescent health and wellbeing. Lancet. 2016 Jun 11;387(10036):2423-78. doi: 10.1016/S0140-6736(16)00579-1. Epub 2016 May 9. No abstract available. PMID 27174304
- [Background] Gottschalk LB, Ortayli N. Interventions to improve adolescents' contraceptive behaviors in low- and middle-income countries: a review of the evidence base. Contraception. 2014 Sep;90(3):211-25. doi: 10.1016/j.contraception.2014.04.017. Epub 2014 May 4. PMID 24916724
- [Background] L'Engle KL, Mangone ER, Parcesepe AM, Agarwal S, Ippoliti NB. Mobile Phone Interventions for Adolescent Sexual and Reproductive Health: A Systematic Review. Pediatrics. 2016 Sep;138(3):e20160884. doi: 10.1542/peds.2016-0884. Epub 2016 Aug 23. PMID 27553221
- [Background] Ministry of Health and Social Welfare (TZ). National Family Planning Guidelines and Standards [Internet]. Dar es Salaam: Ministry of Health and Social Welfare, 2013 [cited 2018 Sept. 19]. 54 p. Available from: https://www.prb.org/wp-content/uploads/2018/05/National-Family-Planning-Guidelines-and-Standards-2013.Tanzania.pdf
- [Background] Agarwal S, LeFevre AE, Lee J, L'Engle K, Mehl G, Sinha C, Labrique A; WHO mHealth Technical Evidence Review Group. Guidelines for reporting of health interventions using mobile phones: mobile health (mHealth) evidence reporting and assessment (mERA) checklist. BMJ. 2016 Mar 17;352:i1174. doi: 10.1136/bmj.i1174. No abstract available. PMID 26988021
- [Background] Bitzer J, Abalos V, Apter D, Martin R, Black A; Global CARE (Contraception: Access, Resources, Education) Group. Targeting factors for change: contraceptive counselling and care of female adolescents. Eur J Contracept Reprod Health Care. 2016 Dec;21(6):417-430. doi: 10.1080/13625187.2016.1237629. Epub 2016 Oct 5. PMID 27701924
- [Background] Cleland J. Illustrative questionnaire for interview-surveys with young people. In: Cleland J, Ingham R, Stone N, eds. Asking Young People About Sexual and Reproductive Behaviors. Illustrative Core Instruments. Geneva: WHO, 2001.
- [Background] Ingham R, Stone N. Topics for In-depth Interviews and Focus Group Discussions: Partner selection, sexual behaviour and risk taking. In: Cleland J, Ingham R, Stone N, eds. Asking young people about sexual and reproductive behaviours: Illustrative Core Instruments. Geneva: WHO, 2001.
- [Background] Ministry of Health, Community Development, Gender, Elderly and Children (TZ). Standard Treatment Guidelines & National Essential Medicines List Tanzania Mainland [Internet]. Dar es Salaam: Ministry of Health, Community Development, Gender, Elderly and Children, 2018 [cited 2018 Sept. 19]. 445 p. Available from: http://www.tzdpg.or.tz/fileadmin/documents/dpg_internal/dpg_working_groups_clusters/cluster_2/health/Key_Sector_Documents/Tanzania_Key_Health_Documents/STANDARD_TREATMENT_GUIDELINES__CORRECT_FINAL_USE_THIS-1.pdf
- [Background] Sexual Reproductive Health and Rights Africa Trust (ZA). Age of Consent: Legal Review Tanzania Country Report [Internet]. Johannesburg: Sexual Reproductive Health and Rights Africa Trust, 2016 [cited 2018 Sept. 19]. 15 p. Available from: https://www.satregional.org/wp-content/uploads/2018/05/Age-of-consent-Tanzania.pdf
- [Background] Johnson D, Juras R, Riley P, Chatterji M, Sloane P, Choi SK, Johns B. A randomized controlled trial of the impact of a family planning mHealth service on knowledge and use of contraception. Contraception. 2017 Jan;95(1):90-97. doi: 10.1016/j.contraception.2016.07.009. Epub 2016 Jul 13. PMID 27421767
- [Background] Vahdat HL, L'Engle KL, Plourde KF, Magaria L, Olawo A. There are some questions you may not ask in a clinic: providing contraception information to young people in Kenya using SMS. Int J Gynaecol Obstet. 2013 Nov;123 Suppl 1:e2-6. doi: 10.1016/j.ijgo.2013.07.009. Epub 2013 Aug 2. PMID 24012514